CLINICAL TRIAL: NCT05624476
Title: Pan-genome Sequencing of Urine Cell-free DNA for Therapy of Urinary Infectious Diseases: a Single Center Prospective Study Clinical Control Study
Brief Title: mNGS for Therapy of Urinary Infectious Diseases
Acronym: PGS-U-UTI&UC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CZGR2022002
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Urinary Tract Infections; Sequelae of; Infection
MeSH Terms: conditions — Urinary Tract Infections; Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — free cfDNA of pathogens in urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: Patients with urinary tract infection received treatments guided by both culture and mNGS
  Interventions: Diagnostic Test: mNGS of urine cell-free DNA
- control group: Patients with urinary tract infection received treatments guided by culture first
  Interventions: Diagnostic Test: mNGS of urine cell-free DNA

INTERVENTIONS:
Diagnostic Test: mNGS of urine cell-free DNA — Metagenomic sequencing of urine cell-free DNA

SUMMARY:
Urinary tract infection is a common infectious disease in clinic. Although urinary tract infection can be initially diagnosed by clinical sign and symptom, signs and urine routine, the application of appropriate antibiotic therapy depends on the further identification of pathogens.

Metagenomic sequencing has been widely used in clinical pathogen diagnosis, especially in difficult infectious diseases. ICompared with tissue samples, cerebrospinal fluid, bronchoalveolar lavage fluid, whole blood and other samples, the application of mNGS in urine samples is relatively limited because incorrect sampling methods before and after collection of urine samples are easy to contaminate the samples and the colonization of distal urethra, periurethral skin and vagina will interfere with the interpretation of reports.

Previous small sample studies have shown that the sensitivity of mNGS in urinary tract infection is high, but the specificity is relatively low, and there are many problems such as difficult interpretation of reports and low clinical conformity. This is closely related to the mNGS technology algorithm, such as the inability to eliminate the influence of urinary system background bacteria, and the ambiguity of short sequence alignment, which makes it difficult to distinguish homologous pathogens.

In this study, based on the standard mNGS sequencing process, the improved Z value analysis method was used to select strictly enrolled clinical samples and compare them with pathogen culture to observe the clinical value of mNGS with Z value analysis method in the treatment of urinary tract infection.

DETAILED DESCRIPTION:
Urinary tract infection is a common infectious disease in clinic. Urinary tract infection is easily caused by abnormal structure and function of urinary system, low immunity, pregnancy, gender and sexual activity, and iatrogenic factors. Urinary tract infection has a wide spectrum of pathogenic microorganisms, including Gram-negative bacilli, Gram-positive cocci, fungi, mycoplasma, chlamydia, viruses and so on. Although urinary tract infection can be initially diagnosed by clinical sign and symptom, signs and urine routine, the application of appropriate antibiotic therapy depends on the further identification of pathogens. At present, it is commonly used to collect midstream urine for pathogen culture in clinic, but it has the disadvantages of time-consuming and low detection rate, and the use of antibiotics can affect the results of culture.

Metagenomic sequencing has been widely used in clinical pathogen diagnosis, especially in difficult infectious diseases. Its principle is to collect samples, use mNGS to process the samples before sequencing, expose the nucleic acid, compare the nucleic acid sequence of pathogens with the designated huge biological database, and realize the comprehensive detection of viruses, bacteria, fungi, parasites and atypical microorganisms. Compared with tissue samples, cerebrospinal fluid, bronchoalveolar lavage fluid, whole blood and other samples, the application of mNGS in urine samples is relatively limited because incorrect sampling methods before and after collection of urine samples are easy to contaminate the samples and the colonization of distal urethra, periurethral skin and vagina will interfere with the interpretation of reports. However, mNGS has obvious advantages in clinical diagnosis, with high specificity and accuracy, and shorter detection time than traditional culture. In the aspect of mixed infection, because of its non-bias, the detection rate of multiple pathogens is higher than that of conventional culture, smear, PCR and other tests, which can detect other pathogens and even rare pathogens that can not be detected conventionally.

Previous small sample studies have shown that the sensitivity of mNGS in urinary tract infection is high, but the specificity is relatively low, and there are many problems such as difficult interpretation of reports and low clinical conformity. For example, there are many pathogens with high reading, and the test results are sorted to form a list of pathogens, but it is impossible to determine which or which pathogens are pathogenic. This is closely related to the mNGS technology algorithm, such as the inability to eliminate the influence of urinary system background bacteria, and the ambiguity of short sequence alignment, which makes it difficult to distinguish homologous pathogens.

In this study, based on the standard mNGS sequencing process, the improved Z value analysis method was used to select strictly enrolled clinical samples and compare them with pathogen culture to observe the clinical value of mNGS with Z value analysis method in the treatment of urinary tract infection.

ELIGIBILITY:
Inclusion Criteria:

* Age: 16-70 years.
* Typical symptoms of urinary tract infection + pyuria (WBC ≥ 10/HP in urine sediment after centrifugation).
* Clinical diagnosis: acute cystitis, urethritis, acute and chronic prostatitis, pyelonephritis, epididymitis; or complex urinary tract infection, such as urinary tract deformity, obstruction, double J tube, etc.
* Sign the informed consent form voluntarily.

Exclusion Criteria:

* Malignant tumors of liver or other organs or previous history of tumors.
* Complicated with gastrointestinal bleeding, spontaneous bacterial peritonitis, hepatic encephalopathy, hepatorenal syndrome and acute infection.
* Patients with severe heart, lung, kidney or blood system diseases and failure.
* Pregnant or breastfeeding women.
* Allergic constitution.
* Those who have a history of alcoholism and drug abuse and fail to give up effectively.
* The subject withdrew from the study on the condition that he/she had not participated in other clinical trials within 4 weeks.
* Other conditions which, in the opinion of the investigator, are not suitable for participation in the study.
* Antibiotic therapy was performed in the past month because of urinary tract infection.
* Broad-spectrum antibiotic therapy has been performed for other uncontrollable infections or other infections.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with urinary tract infection, which is caused by abnormal structure and function of urinary system, low immunity, pregnancy, gender and sexual activity, and iatrogenic factors, with a wide spectrum of pathogenic microorganisms, including Gram-negative bacilli, Gram-positive cocci, fungi, mycoplasma, chlamydia, viruses and so on, and diagnosed by clinical sign and symptom, signs and urine routine.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants cured from urinary tract infection | 17 days
  The "cure" is defined as "The clinical symptom of urinary tract infection disappeared and the urine tests returned to normal"

CONTACTS AND LOCATIONS:
Overall Officials: Junxue Wang, Prof., Principal Investigator — Changzheng Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Flores-Mireles AL, Walker JN, Caparon M, Hultgren SJ. Urinary tract infections: epidemiology, mechanisms of infection and treatment options. Nat Rev Microbiol. 2015 May;13(5):269-84. doi: 10.1038/nrmicro3432. Epub 2015 Apr 8. PMID 25853778
- [Result] Frimodt-Moller N. The urine microbiome - Contamination or a novel paradigm? EBioMedicine. 2019 Jun;44:20-21. doi: 10.1016/j.ebiom.2019.05.016. Epub 2019 May 14. No abstract available. PMID 31101594
- [Result] Janes VA, Matamoros S, Munk P, Clausen PTLC, Koekkoek SM, Koster LAM, Jakobs ME, de Wever B, Visser CE, Aarestrup FM, Lund O, de Jong MD, Bossuyt PMM, Mende DR, Schultsz C. Metagenomic DNA sequencing for semi-quantitative pathogen detection from urine: a prospective, laboratory-based, proof-of-concept study. Lancet Microbe. 2022 Aug;3(8):e588-e597. doi: 10.1016/S2666-5247(22)00088-X. Epub 2022 Jun 7. PMID 35688170
- [Result] Foxman B. Urinary tract infection syndromes: occurrence, recurrence, bacteriology, risk factors, and disease burden. Infect Dis Clin North Am. 2014 Mar;28(1):1-13. doi: 10.1016/j.idc.2013.09.003. Epub 2013 Dec 8. PMID 24484571
- [Result] Mitchell SL, Simner PJ. Next-Generation Sequencing in Clinical Microbiology: Are We There Yet? Clin Lab Med. 2019 Sep;39(3):405-418. doi: 10.1016/j.cll.2019.05.003. PMID 31383265
- [Result] Zeng S, Ying Y, Xing N, Wang B, Qian Z, Zhou Z, Zhang Z, Xu W, Wang H, Dai L, Gao L, Zhou T, Ji J, Xu C. Noninvasive Detection of Urothelial Carcinoma by Cost-effective Low-coverage Whole-genome Sequencing from Urine-Exfoliated Cell DNA. Clin Cancer Res. 2020 Nov 1;26(21):5646-5654. doi: 10.1158/1078-0432.CCR-20-0401. Epub 2020 Oct 9. PMID 33037018